CLINICAL TRIAL: NCT02041728
Title: The Detection of Early Dementia With the Digital Game Memory
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S54845
Record Dates: First submitted 2013-06-26; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators are going to test if it is possible to detect early dementia with the digital game "memory". The investigators are going to test 15 healthy people and 15 patients with early dementia.

The test consists of playing the game "memory" several times. While playing, several parameters are stored.

The investigators are going to test if any correlation can be found between these parameters and the cognitive state of the person as tested by the Mini-Mental status examination.

ELIGIBILITY:
Inclusion Criteria:

* healthy 75-plusser
* 75-plusser with early dementia

Exclusion Criteria:

* younger than 75
* patient with other cognitive impairments than dementia

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: * healthy subjects of 75 or older
  * subjects with mild dementia of 75 or older
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Association of cognitive status with failures in a computerised memory game | The game will be played once during 10-30 minutes.
  Failure is defined as the number of trials for the memory task

CONTACTS AND LOCATIONS:
Overall Officials: Jos Tournoy, Principal Investigator — University of Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium